CLINICAL TRIAL: NCT06912022
Title: Supporting Antibiotic Stewardship in Primary Care Via Point-of-care Testing (POCT) for Acute Respiratory Tract Infections
Brief Title: ASPIRE I: Supporting Antibiotic Stewardship in Primary Care Via POCT
Acronym: ASPIRE I
Status: Completed | Type: Observational
Sponsor: University of South Wales (Other)
Collaborators: Cwm Taf University Health Board (NHS) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 306081
Record Dates: First submitted 2022-02-24; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Acute Respiratory Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspected ARI patients: Patient presenting with acute respiratory infections tested using the FebriDx POC assay.
  Interventions: Device: FebriDx Device

INTERVENTIONS:
Device: FebriDx Device — Patients suspected of an acute respiratory infection were tested using the FebriDx POC assay.

SUMMARY:
The ASPIRE study is an uncontrolled observational feasibility study, and a collaboration between the University of South Wales and Cwm Taf Morgannwg University Health Board (CTMUHB). The study is based at Ysbyty Cwm Rhondda (YCR) and Keir Hardy Primary Care (KHPC) centres, where participant recruitment will take place. Study participants will be invited to provide capillary blood samples (via finger prick sampling) for testing. The principal investigators are Dr Aled Davies at YCR and Dr Shyama Velupillai at KHPC. Upon clinical assessment, and after provision of consent, participants will undergo an ARI (acute respiratory infection) POC assay. This is a dual marker immunoassay designed to detect raised levels of C-reactive protein and MxA in capillary blood. The assay uses the sensitivity of CRP and specify of MxA to aid in the differentiation of ARI's in Primary Care.

The POC assay results will be compared to the participants clinical outcomes and the physician directed treatment pathway via reviewing medical records and by contacting the patient from 14 days after their visit.

DETAILED DESCRIPTION:
Antibiotic stewardship is fast becoming an essential measure to improve antibiotic prescribing by clinicians. Antibiotic stewardship not only presents a cost-effective strategy for the NHS but addressed the issue of antimicrobial resistance (AMR) and protects patients from harm caused by unnecessary antibiotic use.

The economic costs of antibiotic resistance are largely unknown, but it is anticipated that with an increased number of cases, effects to the economy could be severe. Infections and infectious diseases cost England & Wales an estimated £30 billion a year, with many cases of acute respiratory infections (Chaplin, 2017). POC diagnostic tests in a clinical setting could give clinicians the ability to distinguish between microbial and viral infections, providing a more informed decision to antibiotic prescribing.

The purpose of this study is to safely distinguish between bacterial or viral respiratory infections in a primary care setting using "point of care" (POC) testing to provide a retrospective insight as to whether clinical assessment of an acute respiratory infection (ARI) is justified. Upon clinical assessment, the current clinical practice prescribes antibiotics based on symptoms reported by the patient and a subjective review by the GP. This results in antibiotics being prescribed from an informed decision made by the clinician, based only from patient symptoms. The use of a dual marker immunoassay could guide informed decisions based on qualitative data and degree of infection using POC testing in Primary Care.

The POC assay uses a dual marker immunoassay to differentiate between a viral and bacterial infection. C-reactive protein (CRP) is raised in the blood stream in response to inflammation. CRP can be elevated in viral infections, but generally the rise is to higher levels in bacterial infections, especially severe bacterial infections. Another blood protein, the MxA protein, is selectively increased in people with viral infections and therefore has the potential to greatly enhance the rapid distinction between viral and bacterial respiratory infections.

NICE guidance from 2014 recommends the use of CRP POC test in the diagnosis and appropriate management of lower respiratory tract infections in adults aged 18 and over (excluding people with COPD) after clinical assessment whether antibiotics should be prescribed. The study POC assay data could be used as an effective tool alongside NICE guidelines to prescribe antibiotics based on CRP concentration where an infection may be viral. Recent clinical studies suggest the POC test is highly effective, yielding over 80% sensitivity and over 90% specificity when identifying bacterial and viral infections in adults (NICE, 2020).

ELIGIBILITY:
Inclusion Criteria:

* Subject >18 years of age.
* Having new onset symptoms suggestive of acute respiratory infection (ARI within 7 days of seeking care: runny nose, nasal congestion, sore throat, cough, hoarse voice, softness of breath) with or without fever.

Exclusion Criteria:

* Unable to provide informed consent.
* Undergoing end of life care.
* Immunocompromised or taking chemotherapy, oral steroids, or interferon.
* Receiving a live vaccine in the last 14 days.
* Taking antibiotics or antivirals in the last 14 days.
* Patients that are systematically unwell or having symptoms that lasted more than 7 days*.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be recruited from self-referred patients attending YCR and KHPC centres with a self-suspected acute respiratory infection (ARI). The study aims to collect a minimum of 140 participants using a pragmatic sampling regime. The feasibility study will provide the data required to design and conduct a more detailed and statistically powered trial.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Concordance between FebriDx result and Clinician Decision | Feb 2023
  The level of agreement between the FebriDx classification (viral or bacterial) and the clinician's initial diagnostic impression and treatment decision (i.e. prescribe antibiotics or not).

SECONDARY OUTCOMES:
Sensitivity and Specificity of FebriDx vs.Clinical Judgement | Feb 2023
  Sensitivity (true positive rate) and specificity (true negative rate) of FebriDx in identifying bacterial or viral infections, using clinical decision as reference.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Mark Williams, PhD, Study Director — Chief Investigator University of South Wales
Locations (2):
- United Kingdom (2):
  - Keir Hardie Practice 3, Cardiff
  - Ysbyty Cwm Rhondda, Cardiff

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/22/NCT06912022/Prot_000.pdf